CLINICAL TRIAL: NCT06785623
Title: Improvement of Depression in Terminal Cancer Patients (IDTCP)
Brief Title: Improvement of Depression in Terminal Cancer Patients
Acronym: IDTCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202409106RIND
Record Dates: First submitted 2025-01-06; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-12

CONDITIONS: Depression; Cancer Patients and Depression and Suicide; Life Quality
Keywords: depression; terminal cancer patients; palliative care
MeSH Terms: conditions — Depression; Suicide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastrodia elata Blume water extract (Experimental): Subjects will receive Gastrodia elata Blume water extract
  Interventions: Dietary Supplement: Gastrodia elata Blume water extract
- Gastrodia elata Blume water extract-like (Placebo Comparator): Subjects will receive a placebo resembling Gastrodia elata Blume water extract
  Interventions: Dietary Supplement: Gastrodia elata Blume water extract

INTERVENTIONS:
Dietary Supplement: Gastrodia elata Blume water extract — Subjects in the experimental group will consume Gastrodia elata Blume water extract daily. The extract is prepared from dried Gastrodia elata Blume, which is processed into a water-soluble form. This dosage is administered orally for a duration of a week. The intervention is designed to evaluate the potential effects of Gastrodia elata Blume on alleviating depressive symptoms, improving autonomic nervous system function, and enhancing overall quality of life in terminal cancer patients.

SUMMARY:
This study investigates the potential of the water extract of Gastrodia elata Blume (WGE) to alleviate depressive symptoms in terminal cancer patients. In Taiwan, cancer accounts for 25-30% of annual deaths, with terminal patients often experiencing physical pain and psychological distress, including depression. Addressing both physical and psychological challenges is vital in palliative care.

Gastrodia elata Blume is a traditional dietary medicine known for its antidepressant, anti-inflammatory, antioxidant, neurotransmitter-regulating, and neuroprotective properties. This trial will recruit 60 hospice patients, randomly divided into two groups: a control group and a WGE experimental group.

Assessments will include:

1. General examinations (e.g., height, weight, blood pressure).
2. Non-invasive autonomic nervous system analyses.
3. Patient-reported measures: Quality of Life Scale (EORTC QLQ-C30), Pain Score, and Hospital Anxiety and Depression Scale (HADS).

The study hypothesizes that WGE can:

1. Alleviate depressive symptoms.
2. Enhance autonomic nervous system function.
3. Improve the quality of life for terminal cancer patients.

This research aims to demonstrate the therapeutic potential of WGE, improving psychological and physiological outcomes for hospice patients.

DETAILED DESCRIPTION:
In Taiwan, the annual number of cancer-related deaths constitutes approximately 25-30% of the overall mortality rate. Terminal cancer patients often endure physical pain and psychological distress, leading to varying degrees of depression. Aligning with the objectives of palliative care, it is crucial to address both the physical pain and psychological well-being of patients. Gastrodia elata Blume (GE), a key component in traditional dietary medicine, has been extensively studied for its diverse biological activities, including antidepressant effects, anti-inflammatory properties, antioxidant capabilities, neurotransmitter regulation, and neuroprotection. This study aims to harness the antidepressant properties of GE to alleviate depression among hospice patients. The trial plans to recruit 60 subjects from the hospice ward, randomly assigning them to either a non-GE group or a GE experimental group (where subjects will consume water extract from 8 g of dried GE daily). Prior to and post each assessment, medical professionals will conduct general examinations (height, weight, blood pressure) and non-invasive autonomic nervous system analyses. Additionally, subjects will complete the Quality of Life Scale (EORTC QLQ-C30), Pain Score, and Hospital Anxiety and Depression Scale (HADS) to facilitate subsequent statistical analysis and evaluate the antidepressant efficacy of GE water extract. This experiment aims to demonstrate that GE water extract can improve depression in hospice patients, enhancing their autonomic nervous system function and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years
* Diagnosis of terminal cancer, with an expected life expectancy of less than 6 months-
* Patients with sufficient cognitive status to respond to the research staff's evaluation questions

Exclusion Criteria:

* Patients or their families who refuse to participate
* Patients who withdraw from the study
* Patients who have participated in other research studies within one month before or during the trial
* Patients with suicidal tendencies

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-14 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in Depressive Symptoms | 1 week
  Hospital Anxiety and Depression Scale (HADS)
  Outcome Measure Title: Hospital Anxiety and Depression Scale (HADS) Total Score Description: The HADS is a 14-item questionnaire used to measure anxiety and depression levels in participants. Each item is scored on a 4-point Likert scale ranging from 0 to 3, with separate scores calculated for the Anxiety subscale (HADS-A) and Depression subscale (HADS-D).
  Minimum Score: 0 Maximum Score: 21 per subscale (42 total for both subscales combined) Interpretation: Higher scores indicate worse outcomes (greater severity of anxiety or depression).
Improvement in Quality of Life | 1 week
  European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
  Outcome Measure Title: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Description: The EORTC QLQ-C30 is a 30-item questionnaire designed to assess the quality of life of cancer patients. It includes multi-item scales that evaluate global health status, functional domains (physical, role, emotional, cognitive, and social functioning), and symptom scales (e.g., fatigue, pain, nausea/vomiting).
  Minimum Score: 0 Maximum Score: 100 for each scale (scores are linearly transformed to a 0-100 scale).
  Interpretation: For global health status and functional scales, higher scores indicate better outcomes (better functioning or quality of life). For symptom scales, higher scores indicate worse outcomes (greater symptom burden).
Changes in Pain Score | 1 week
  pain score
  Outcome Measure Title:Pain Intensity Measurement Using the Numeric Pain Rating Scale (NPRS) Description of the Measurement Tool:The Numeric Pain Rating Scale (NPRS) is a self-reported measure commonly used to assess pain intensity. It asks participants to rate their pain on a scale from 0 (No Pain) to 10 (Worst Pain Possible). The scale is visualized using smiley faces, transitioning from green (mild/no pain) to red (severe pain).
  Scoring Details:
  Minimum Value: 0 (indicating no pain). Maximum Value: 10 (indicating the worst pain possible).
  Interpretation:
  Higher scores indicate worse outcomes (i.e., more severe pain). Lower scores indicate better outcomes (i.e., less or no pain).
Changes in heart rate variability | 1 week
  Heart Rate Monitor (GSH751) is a non-invasive device approved by Taiwan's Ministry of Health (Certification No. 006983). It measures heart rate through finger electrodes and uses Bluetooth to transmit data for recording and analysis. The device evaluates heart rate variability (HRV) and autonomic nervous system function, including parameters like heart rate, SDNN (autonomic health indicator), sympathetic (LF), parasympathetic (HF) activity, and LF/HF balance index. Time domain and frequency domain analyses help assess stress, anxiety, sleep disorders, and overall autonomic balance, enabling users to track long-term health trends.
  (Model: GSH751, Approved by Taiwan Ministry of Health, Certification No. 006983)

CONTACTS AND LOCATIONS:
Overall Officials: Jaw Shiun Tsai, Study Chair — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No